CLINICAL TRIAL: NCT06044805
Title: Monitoring Therapeutic Efficacy of Chloroquine Plus Primaquine in the Treatment of Uncomplicated Plasmodium Vivax Based on Clinical, Parasitologic and Hematologic Parameters in Shecha Health Center: Open Label Clinical Trial
Brief Title: Therapeutic Efficacy of Chloroquine Plus Primaquine in the Treatment of Uncomplicated Plasmodium Vivax
Acronym: CQ+PQ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dinka Dugassa (Other)
Collaborators: Ethiopian Public Health Institute (Other Government)
Responsible Party: Sponsor-Investigator, Dinka Dugassa, Principal Investigator, Wollega University
Organization: Wollega University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPHI-IRB-294-2
Record Dates: First submitted 2023-07-06; First posted 2023-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Efficacy; Malaria; Chloroquine; Vivax Malaria
Keywords: Therapeutic; Efficacy; Chloroquine; Primaquine; Ethiopia
MeSH Terms: conditions — Malaria; Malaria, Vivax | interventions — Chloroquine; chloroquine diphosphate; Primaquine

STUDY DESIGN:
Intervention Model Description: Open label clinical trial study will be conducted in Shecha Health Center from December 2022 to March 2023. Participants will be selected and treated with a 25 mg/kg standard dose of chloroquine over three days and a 0.25 mg/kg standard dose of primaquine over fourteen days. Clinical, parasitologic, and hematologic parameters will be monitored for up to a 42-day follow-up period, which will be used to evaluate therapeutic efficacy of CQ+PQ. Thick and thin blood smears will be prepared and examined to determine parasite clearance, and clinical examination will be performed over 42 follow up periods. Haemoglobin level will be measured on days 0, 14, 28 and 42. WHO double-entry Excel sheet will be used for KaplanMeier survival analysis and SPSS version-26 software will be used to analyse the data. All comparisons will be performed at 95% confidence interval and a significance level of 0.05, Pvalue of <0.05 will be considered statistically significant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic Efficacy of Chloroquine Plus Primaquine (Experimental): An invivo single arm trial. Chloroquine (tablet containing 150mg of base) - it was given on days 0 (10mg/kg), 1(10mg/kg) and 2 (5mg/kg). Total dose, 25 mg base/kg.
  Primaquine - it was given once a day (0.25 mg/kg) for fourteen days, starting on day 0 of CQ treatment. Total dose, 3.5mg/kg.
  The medications were administered under direct observation and the patient was monitored for vomiting for 60 minutes.
  Interventions: Drug: Chloroquine; Drug: Primaquine

INTERVENTIONS:
Drug: Chloroquine — Total of 25mg base per kg over 3 days (10 mg base/kg on Days 0 and 1, 5 mg base/kg on Day 2)
  Other Names: Chloroquine base; Chloroquine Phosphate
Drug: Primaquine — Primaquine: 7.5 mg base tablet. Medication given as 0.25mg/kg daily for 14 days.

SUMMARY:
The goal of this open label clinical trial will be to assess the therapeutic efficacy of chloroquine plus primaquine in the treatment of uncomplicated plasmodium vivax in Shecha Health Center, South Ethiopia.

The main question it aims to answer:- the current therapeutic efficacy of chloroquine plus primaquine in the treatment of uncomplicated plasmodium vivax in Shecha Health Center, South Ethiopia based on clinical, parasitological and hematological parameter.

Participants will be patients aged >6 months with diagnosis of plasmodium vivax mono-infection and who fulfills the inclusion criteria.

This is a single arm open label invivo therapeutic efficacy study of chloroquine plus primaquine in the treatment of uncomplicated plasmodium vivax. The final result will be compared with World Health Organization recommendation on antimalarial drug therapeutic efficacy.

DETAILED DESCRIPTION:
The goal of this open label clinical trial will be to assess the therapeutic efficacy of chloroquine plus primaquine in the treatment of uncomplicated plasmodium vivax in Shecha Health Center, South Ethiopia. The main question it aims to answer:- the current therapeutic efficacy of chloroquine plus primaquine in the treatment of uncomplicated plasmodium vivax in Shecha Health Center, South Ethiopia based on clinical, parasitological and hematological parameter.

Participants will be patients aged >6 months with diagnosis of plasmodium vivax mono-infection and who fulfills the inclusion criteria.

This is a single arm open label invivo therapeutic efficacy study of chloroquine plus primaquine in the treatment of uncomplicated plasmodium vivax. The final result will be compared with World Health Organization recommendation on antimalarial drug therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 6 months
* Slide confirmed infection with P. vivax with > 250 asexual forms/μl
* Lives within 5 km of the enrolling health facility
* Weight ≥ 5.0 kg
* Ability to swallow oral medication
* Ability and willingness to comply with the protocol for the duration of the study and to comply with the study visit schedule
* Informed consent from patient or from a parent or guardian in the case of children

Exclusion Criteria:

* Sever malaria with complication sign and symptoms
* Signs or symptoms of severe malnutrition, defined as weight-for-age ≤ 3 standard deviations below the mean, symmetrical edema involving at least the feet, or mid-upper arm circumference <100 cm for children less than five years of age
* Mixed plasmodium infection
* Severe anemia, defined as hemoglobin (Hb) < 5 g/dl
* Presence of febrile conditions caused by diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhea with dehydration)
* Serious or chronic medical condition (e.g. cardiac, renal, hepatic diseases, sickle cell disease, HIV/AIDS)
* Positive pregnancy test or breastfeeding
* Unable or unwilling to take contraceptives for women of child-bearing age
* Children weighing less than 5 kilograms
* History of hypersensitivity reaction to any medication tested or used as an alternative treatment
* Participants with history of prolonged QT conditions
* Taking regular medication, which may interfere with antimalarial pharmacokinetics or efficacy

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Early treatment failure [Time Frame: within the first 3 days] | within the first 3 days
  Danger signs or severe malaria on day 1, day 2 or day 3 in the presence of parasitemia;Parasitemia on day 2 higher than on day 0, irrespective of axillary temperature;Parasitemia on day 3 with axillary temperature ≥37.5 ºC;Parasitemia on day 3 ≥25% of count on day 0.
Late Clinical Failure (LCF) | 42 days
  Danger signs or severe malaria in the presence of parasitemia on any day between day 4 and 42 in patients who did not previously meet any of the criteria of Early Treatment Failure; Presence of parasitemia on any day between 4 and day 42 with axillary temperature ≥37.5 °C (or history of fever) in patients who did not previously meet any of the criteria of Early Treatment Failure.
Late Parasitological Failure (LPF) | 42 days
  Presence of parasitemia on any day between day 7 and day 42 and axillary temperature <37.5 ºC in patients who did not previous meeting any of the criteria of Early Treatment Failure or Late Clinical Failure.
Adequate Clinical and Parasitological Response (ACPR) | 42 days
  Absence of parasitemia on day 42 irrespective of axillary temperature, in patients who did not previously meet any of the criteria of Early Treatment Failure, Late Clinical Failure, or Late Parasitological Failure.

SECONDARY OUTCOMES:
The secondary outcome of this study is determining parasite clearance rate based on parasite clearance time. | 42 days
  This study's secondary goal was to calculate the parasite clearance rate based on parasite clearance time. Using hours, days, weeks, and months, parasite clearance time is calculated.
The secondary outcome of this study is determining gametocyte clearance rate based on gametocyte clearance time. | 42 days
  This study's secondary goal was to calculate the gametocyte clearance rate based on gametocyte clearance time. Using hours, days, weeks, and months, parasite clearance time is calculated.
The secondary outcome of this study is determining fever clearance rate based on fever clearance time. | 42 days
  Calculating the fever clearance rate based on fever clearance time was the secondary outcome of this clinical trial. Fever clearance time is calculated using hours, days, weeks, and months. Temperatures less than 37.5 degrees celsius (T 37.5oC) are deemed to be fever-free(fever cleared) while temperatures greater than or equal to 37.5 degrees celsius (T>37.5oC) are classified as having fever (fever not cleared).
The secondary outcome of this study is determining mean hemoglobin change overtime in the 42 days study period. | 42 days
  Calculating the mean hemoglobin change overtime in the 42 study period based on hemoglobin concentration at D0, D14, D28 and D42 was the secondary outcome of this clinical trial. Milligrammes per deciliter are used to measure the concentration of haemoglobin.
The secondary outcome of this study is evaluating the incidence of adverse events in 42 follow-up period. | 42 days
  This study's secondary goal was evaluating the incidence of adverse events in 42 follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Bockretsion Gidey, Study Director — Ethiopian Public Health Institute
Locations (1):
- Shecha Health Center, Arba Minch, South Ethiopia, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fekadu G, Dugassa D, Negera GZ, Woyessa TB, Turi E, Tolossa T, Fetensa G, Assefa L, Getachew M, Shibiru T. Self-Medication Practices and Associated Factors Among Health-Care Professionals in Selected Hospitals of Western Ethiopia. Patient Prefer Adherence. 2020 Feb 20;14:353-361. doi: 10.2147/PPA.S244163. eCollection 2020. PMID 32110001
- [Result] Fekadu G, Bekele F, Tolossa T, Fetensa G, Turi E, Getachew M, Abdisa E, Assefa L, Afeta M, Demisew W, Dugassa D, Diriba DC, Labata BG. Impact of COVID-19 pandemic on chronic diseases care follow-up and current perspectives in low resource settings: a narrative review. Int J Physiol Pathophysiol Pharmacol. 2021 Jun 15;13(3):86-93. eCollection 2021. PMID 34336132
- [Result] Bekele F, Fekadu G, Bekele K, Dugassa D, Sori J. Drug-related problems among patients with infectious disease admitted to medical wards of Wollega University Referral Hospital: Prospective observational study. SAGE Open Med. 2021 Jan 22;9:2050312121989625. doi: 10.1177/2050312121989625. eCollection 2021. PMID 33552517
- [Result] Fekadu G, Turi E, Kasu T, Bekele F, Chelkeba L, Tolossa T, Labata BG, Dugassa D, Fetensa G, Diriba DC. Impact of HIV status and predictors of successful treatment outcomes among tuberculosis patients: A six-year retrospective cohort study. Ann Med Surg (Lond). 2020 Nov 15;60:531-541. doi: 10.1016/j.amsu.2020.11.032. eCollection 2020 Dec. PMID 33299558

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT06044805/Prot_SAP_ICF_000.pdf